CLINICAL TRIAL: NCT02505282
Title: Vitamin K Status and Markers of Vascular Function in Patients With and Without Postural Hypotension
Acronym: VITKOH
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Collaborators: British Geriatrics Society (Other)
Responsible Party: Principal Investigator, Matthew Lambert, Clinical Lecturer, University of Dundee
Other Study IDs: 2011CV14
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Orthostatic Hypotension
Keywords: Orthostatic hypotension; Vitamin K
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Orthostatic Hypotension: >20mmHg systolic BP drop or >10mmHg diastolic BP drop on standing, and syncopal symptoms on standing
  Interventions: Other: Vitamin K status
- Control: No fall in BP or <20mmHg systolic BP drop and <10mmHg diastolic BP drop on standing, and no syncopal symptoms on standing
  Interventions: Other: Vitamin K status

INTERVENTIONS:
Other: Vitamin K status — Vitamin K status indicated by desphospho-uncarboxylated matrix Gla protein level

SUMMARY:
Postural hypotension is common in older people, leading to falls, decline in function, and dependence. Available treatments have limited efficacy and tolerability; novel approaches to treatment are therefore needed. Decreased vascular health, stiffening of the arteries and consequent decreased vascular reactivity are thought to contribute to postural hypotension and are therefore therapeutic targets.

Recent trial evidence has suggested that vitamin K may exert beneficial effects on vascular health particularly in respect to inhibiting calcification. Calcification increases vascular stiffness, decreases compliance and thus decreases the ability of blood vessels to autoregulate blood pressure and flow - which could contribute to postural drops in blood pressure. Worsened vascular health could also impact adversely on baroceptor function, which is needed for blood pressure autoregulation and which is disrupted in patients with orthostatic hypotension.

Vitamin K intake is below recommended daily intake in 60% of adults in the UK. In animals, vitamin K supplementation may be able to reverse calcification of arteries, and in humans Vitamin K has been shown to arrest decline in carotid artery elasticity compared to placebo. High levels of circulating vitamin K were also associated with lower levels of CRP in the Framingham cohort, suggesting a possible role in the suppression of chronic inflammation that is known to accompany vascular disease. The recent ECKO study suggested that vitamin K may reduce falls and fractures; an intriguing question that follows on from this is whether this could be due to beneficial effects on vascular health and postural hypotension, leading to less dizziness and reduced falls.

This cross-sectional comparative study aims to find whether there is a difference in the vitamin K status of patients with postural hypotension compared to those without postural hypotension and whether differences in vitamin K status are associated with other markers of vascular function in patients with and without postural hypotension. This could potentially lead to new treatments for the condition for which there is currently little of proven benefit.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* For postural hypotension group: >20mmHg systolic BP drop or >10mmHg diastolic BP drop on standing, and syncopal symptoms on standing.
* For control group: no fall in BP or <20mmHg systolic BP drop and <10mmHg diastolic BP drop on standing, and no syncopal symptoms on standing. No previous diagnosis of orthostatic hypotension.

Exclusion Criteria:

* On warfarin
* Unable to consent
* Unable to stand unaided

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Aged 65 years or older, not on warfarin, able to stand unaided, able to give informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2012-04; Primary Completion 2014-01 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Serum non-phosphorylated, non-carboxylated Matrix Gla Protein | Day 1

SECONDARY OUTCOMES:
Vitamin K1 Level | Day 1
Vitamin D | Day 1
Flow mediated dilatation | Day 1
  Measure of endothelial function
Pulse wave velocity | Day 1
  Measure of arterial stiffness and reflectivity
Carotid intima media thickness | Day 1
Pulse wave augmentation index | Day 1
  Measure of arterial stiffness and refelctivity

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Dundee, Dundee, Angus, United Kingdom